CLINICAL TRIAL: NCT05707052
Title: Comparative Effects of Neck-Trunk Stabilization Exercises and Bobath Therapy on Trunk Control and Upper Limb Function in Children With Spastic Diplegic Cerebral Palsy: A Randomized Clinical Trial
Brief Title: Neck-Trunk Stabilization Exercises and Bobath Therapy Spastic Diplegic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0230
Record Dates: First submitted 2023-01-22; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Cerebral Palsy Spastic Diplegia
Keywords: Bobath; Cerebral palsy; Neck-Trunk Stabilization;
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neck-Trunk Stabilization exercises (Experimental): First neck and trunk exercise involved lifting the head in a modified bridge exercise position so that lower abdominal muscles contracted when the neck was bent, thereby activating the neck flexor muscle and the lower abdominal muscles simultaneously. Second exercise involved pushing the neck backward in supine position to activate the erector muscles of the neck and the upper thoracic vertebrae through the extension of the muscles of the back of the neck. Third exercise activated the deep abdominal muscles in bridge exercise positions so that the participants would experience the posterior inclined movement of the pelvis. Keep each posture for 10 seconds at a time and repeat 10 times with a rest interval of 3 seconds per each.
  Interventions: Other: Neck-Trunk Stabilization Exercises and conventional physical therapy
- Bobath Therapy (Experimental): 1. trunk-pelvic-hip neutral alignment with anterior-posterior weight shifts on the ball,
  2. bilateral upper extremity abduction-traction for lateral weight shift,
  3. prone extension on the ball,
  4. forward weight shift for the trunk and hip extension and forward protective extension,
  5. diagonal weight shifts in flexion-rotation direction,
  6. lateral weight shift for simultaneous activation of flexors and extensors,
  7. bilateral shoulder flexion for latissimus dorsi elongation,
  8. pectoral elongation exercise for trunk extension,
  9. preparatory trunk activities (with continuous and/or intermittent compression and intermittent support),
  10. positioning and holding of the head-trunk Keep each posture for 10 seconds at a time with a rest interval of 3 seconds per each.
  Interventions: Other: Bobath Therapy and conventional physical therapy

INTERVENTIONS:
Other: Neck-Trunk Stabilization Exercises and conventional physical therapy — Neck-Trunk Stabilization Exercises along with conventional physical therapy in which stretching, strengthening, ROMs positioning and electrical stimulation are included.
  Arms: Neck-Trunk Stabilization exercises
Other: Bobath Therapy and conventional physical therapy — Bobath based exercises along with conventional physical therapy in which stretching, strengthening, ROMs positioning and electrical stimulation are included.
  Arms: Bobath Therapy

SUMMARY:
Physiotherapy is widely used in the treatment of children with cerebral palsy. This study is conducted to identify the most appropriate physiotherapy approach. The purpose of the study is to compare two physical rehabilitation strategies i.e., Neck-trunk stabilization exercises and Bobath therapy, to investigate their effectiveness on trunk control and upper limb function. The aims of treatment are to influence muscle tone and improve postural alignment by specific handling technique.

DETAILED DESCRIPTION:
The study will be a Randomized Clinical Trial conducted at the physiotherapy outpatient clinic of the tertiary care hospital in Sialkot, Idrees Hospital. Following the approval of the BASR, the study will be completed within six months. The sample will be taken using a non-probability convenient sampling technique, and the sample will be randomly divided into two groups. A sample size of 44 patients will be taken in this study. There will be two groups. Both groups will receive conventional therapy consisting of stretching, strengthening, range-of-motion exercises, positioning, and electrical stimulation. Group A: This group will receive Neck-Trunk Stabilization exercises. Group B: This group will receive Bobath therapy. The total intervention protocol will be given for six weeks' duration, with three sessions per week of about 45 minutes each. Outcome measures tools will be Segmental Assessment of Trunk Control (SATCo) and Manual Ability Classification System (MACS). Children with spastic diplegic cerebral palsy will be measured at baseline and after 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with spastic diplegic cerebral palsy
* Children with score of GMFCS [2] [3] [4] levels(2, 16).
* Signed consent form from parents/guardians.

Exclusion Criteria:

* Children with visual impairments
* Children with major auditory impairments
* Children with previous orthopedic surgery and Botulium toxin-A injection at least for 6 months
* Children having pharmacological intervention for the inhibition of spasticity
* Contractures
* Uncontrolled seizures
* Focal spasticity

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-03-22 (Estimated)

PRIMARY OUTCOMES:
Segmental Assessment of Trunk Control (SATCo) | 4th week
  Changes from baseline SATCo provides a systematic method of assessing discrete levels of trunk control in children with motor disabilities. The SATCo determines the topmost (most cephalo) segment at which control of the upright posture is poor or not demonstrated i.e. is currently being learned for each of static, active and reactive control.
Manual Ability Classification System (MACS) | 4th week
  Changes from baseline MACS as been used to classify how children with cerebral palsy use their hands when handling objects in daily activities.it is designed to reflect the typical manual performance of child. The ability of children from 4 - 18 years old with cerebral palsy to handle objects in everyday activities can be categorized into 5 levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Raza, MS(OMPT), Principal Investigator — Riphah International University
Locations (1):
- Idrees Hospital, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ejraei N, Ozer AY, Aydogdu O, Turkdogan D, Polat MG. The effect of neck-trunk stabilization exercises in cerebral palsy: randomized controlled trial. Minerva Pediatr (Torino). 2021 Sep 30. doi: 10.23736/S2724-5276.21.06206-6. Online ahead of print. PMID 34590804
- [Background] Acar G, Ejraei N, Turkdogan D, Enver N, Ozturk G, Aktas G. The Effects of Neurodevelopmental Therapy on Feeding and Swallowing Activities in Children with Cerebral Palsy. Dysphagia. 2022 Aug;37(4):800-811. doi: 10.1007/s00455-021-10329-w. Epub 2021 Jun 25. PMID 34173063
- [Background] Desouzart G. Physiotherapy intervention according to the Bobath concept in a clinical case of cerebral palsy. Ortho Res Online J. 2018;3(4).
- [Background] Shin JW, Song GB, Ko J. The effects of neck and trunk stabilization exercises on cerebral palsy children's static and dynamic trunk balance: case series. J Phys Ther Sci. 2017 Apr;29(4):771-774. doi: 10.1589/jpts.29.771. Epub 2017 Apr 20. PMID 28533628
- [Background] Shin JW, Song GB. The effects of neck and trunk stabilization exercises on upper limb and visuoperceptual function in children with cerebral palsy. J Phys Ther Sci. 2016 Nov;28(11):3232-3235. doi: 10.1589/jpts.28.3232. Epub 2016 Nov 29. PMID 27942155